CLINICAL TRIAL: NCT00941421
Title: "Comparision of Diagnostic Value of Oesophagal Videocapsul (VCO) and Oeso-gastro-duodenal Fiber Endoscopy (OGDFE) for the Screening of Oesophagal Varix (OV) for Cirrhotic Patients
Brief Title: Value of Oesophagal Videocapsul and Oeso-gastro-duodenal Fiber Endoscopy for the Screening of Oesophagal Varix for Cirrhotic Patients
Acronym: VCO-VO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD 09/5-G
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Cirrhotic Patient With Suspicion of Portal Hypertension and in a OV Screening Context

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- videocapsul and OGDFE (Other): Each patient have a Fiberoptic endoscopy by videocapsul, followed by one traditional oeso-gastro-duodenal fiberoptic endoscopy
  Interventions: Device: oesophagal videocapsule and oeso-gastro-duodenal fiberoptic endoscopy

INTERVENTIONS:
Device: oesophagal videocapsule and oeso-gastro-duodenal fiberoptic endoscopy — each patient receive one OVC and one OGDFE the same day

SUMMARY:
The purpose of this study is to determine the equivalence or not of diagnosis ability of oesophagal videocapsul versus oeso-gastro-duodenal fiber endoscopy in the screening of oesophagal varix.

ELIGIBILITY:
Inclusion Criteria:

* 18< age< 80
* Diagnosis of a cirrhosis
* suspicion of portal hypertension without known diagnosis of a cirrhosis
* Able to give an inform consent

Exclusion Criteria:

Related to pouplation

* case history of cancer or oesophagal surgery
* case history of an ORL cancer
* case history of evolutive cancer

Related to pathology

* Previous fiberoptic endoscopy with OV diagnosis
* Less than 6 month since last fiberoptic endoscopy

Related to tested device

* clinical suspicion of oesophagal stenosis for a patient presenting a dysphagia to solids
* Zenker diverticuls attested
* clinical suspicion of small intestinal stenosis
* patient with pace-maker or any other inter device
* pregnant women
* deglutition troubles withfalse passage and/or conscience troubles

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Presence or not of oesophagal varix | each fiberoptic endoscopy

SECONDARY OUTCOMES:
Presence of OV with red signs | each exam
Presence of big VO or VO with red signs diagnosed by the two exams | each patient
Discrimination threshold for OV prediction | each exam
analogical visual scale for tolerance of each exam | 30 days after last exam

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU Angers, Angers
  - CH Avicenne, Bobigny
  - CH Beaujon, Clichy
  - CH Saint Philibert, Lomme
  - CH Lyon - Herriot, Lyon
  - Hôpital la conception, Marseille
  - CHU Nantes, Nantes
  - CH Cochin, Paris
  - CHU Bordeaux, Pessac
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse - Purpan, Toulouse

REFERENCES:
- [Derived] Cales P, Sacher-Huvelin S, Valla D, Bureau C, Olivier A, Oberti F, Boursier J, Galmiche JP; multicenter group VO-VCO. Large oesophageal varice screening by a sequential algorithm using a cirrhosis blood test and optionally capsule endoscopy. Liver Int. 2018 Jan;38(1):84-93. doi: 10.1111/liv.13497. Epub 2017 Jul 7. PMID 28622450
- [Derived] Sacher-Huvelin S, Cales P, Bureau C, Valla D, Vinel JP, Duburque C, Attar A, Archambeaud I, Benamouzig R, Gaudric M, Luet D, Couzigou P, Planche L, Galmiche JP, Coron E. Screening of esophageal varices by esophageal capsule endoscopy: results of a French multicenter prospective study. Endoscopy. 2015 Jun;47(6):486-92. doi: 10.1055/s-0034-1391393. Epub 2015 Mar 2. PMID 25730284